CLINICAL TRIAL: NCT01892189
Title: A Randomized, Investigator and Subject-Blind, Placebo-Controlled, Single-Dose, 3-Period, Incomplete Block Cross-Over Study to Evaluate the Effects of Single Oral Administration of TAK-063 on Preventing Ketamine-Induced Brain Activity Changes as Well as Psychotic-Like Symptoms in Healthy Male Adults
Brief Title: Effects of TAK-063 on Preventing Ketamine-Induced Brain Activity Changes as Well as Psychotic-Like Symptoms in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TAK-063_102; U1111-1141-2177 (Other: World Health Organization)
Record Dates: First submitted 2013-06-20; First posted 2013-07-04 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Ketamine-Induced Brain Activity Changes; Psychotic-like Symptoms
Keywords: Drug therapy
MeSH Terms: interventions — Ketamine; 1-(2-fluoro-4-(1H-pyrazol-1-yl)phenyl)-5-methoxy-3-(1-phenyl-1H-pyrazol-5-yl)pyridazin-4(1H)-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Sequence 1: Placebo + TAK-063 3 mg + TAK-063 30 mg (Experimental): Period 1, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 3 milligram (mg), orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 30 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period.
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 2: TAK-063 3 mg + TAK-063 30 mg + Placebo (Experimental): Period 1, Day 1: TAK-063 3 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 30 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period.
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 3: TAK-063 30 mg + Placebo + TAK-063 3 mg (Experimental): Period 1, Day 1: TAK-063 30 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 3 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period.
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 4: Placebo + TAK-063 3 mg + TAK-063 300 mg (Experimental): Period 1, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 3 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period.
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 5: TAK-063 3 mg + TAK-063 300 mg+ Placebo (Experimental): Period 1, Day 1: TAK-063 3 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 6: TAK-063 300 mg + Placebo + TAK-063 3 mg (Experimental): Period 1, Day 1: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 3 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period.
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 7: Placebo + TAK-063 30 mg + TAK-063 300 mg (Experimental): Period 1, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight:
  Period 2, Day 1: TAK-063 30 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 8: TAK-063 30 mg + TAK-063 300 mg + Placebo (Experimental): Period 1, Day 1: TAK-063 30 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight.
  Period 1 & 2 are followed by 7 day washout period.
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo
- Sequence 9: TAK-063 300 mg + Placebo + TAK-063 30 mg (Experimental): Period 1, Day 1: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 2, Day 1: TAK-063 placebo-matching tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight; Period 3, Day 1: TAK-063 30 mg tablets, orally, single dose and ketamine, intravenous administration according to a bolus infusion adjusted to the participant's weight. Period 1 & 2 are followed by 7 day washout period
  Interventions: Drug: Ketamine; Drug: TAK-063; Drug: TAK-063 Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine intravenous administration.
  Other Names: Ketalar™
Drug: TAK-063 — TAK-063 tablets
Drug: TAK-063 Placebo — TAK-063 placebo-matching tablets

SUMMARY:
The purpose of this study is to determine whether ketamine-induced brain activity changes are modulated by TAK-063 administration using neuroimaging battery tests.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-063. This study will look at brain activity changes and treatment of psychotic-like symptoms induced by ketamine, in people who take TAK-063.

The study will enroll approximately 27 participants. Participants will be randomly assigned to one of treatment sequences-which will remain undisclosed to the participants during the study (unless there is an urgent medical need). Participants will receive the following study medications by the end of the study:

* Ketamine intravenous infusion (IV) AND
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient AND
* Two doses of TAK-063 at one of three dose levels All participants will be asked to take 3 tablets and will receive a ketamine IV on the first day of 3 separate study periods. Participants will then be assessed for brain activity changes and other symptoms. This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 7 weeks. Participants will make 6 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy adult male.
4. Speaks English as their first language.
5. Is aged 18 to 45 years, inclusive, at the time of informed consent and first dose of study drug.
6. Weighs at least 50 kg and has a body mass index (BMI) between 18 and 32 kilogram per metre square (kg/m^2), inclusive at Screening.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
8. Has a normal magnetic resonance imaging (MRI) scan and electroencephalogram (EEG) measurement at Screening.

Exclusion Criteria:

1. Has received any investigational compound or ketamine within 30 days prior to Day 1 of Period 1.
2. Has received TAK-063 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality (including MRI or EEG), which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of TAK-063 or ketamine.
6. Has a contraindication for ketamine.
7. Has a positive result for drugs or alcohol at Screening or Check-in (Day -1 of Period 1).
8. Has a history of drug or alcohol abuse or dependence (as defined by Diagnostic & Statistical Manual of Mental Disorders, fourth Edition [DSM-IV]) within 1 year prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
9. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products.
10. Has evidence of current cardiovascular, central nervous system (CNS), hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-063 or ketamine or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
11. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [e.g., cholecystectomy]).
12. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1 of Period 1.
13. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), or a known history of human immunodeficiency virus infection at Screening.
14. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1 of Period 1) or cotinine test is positive at Screening or Check-in (Day -1 of Period 1).
15. Has poor peripheral arterial/venous access or recent wrist trauma.
16. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 3 months prior to Day 1 of Period 1.
17. Has a Screening and/or Check-in (Day -1 of Period 1) abnormal (clinically significant) electrocardiogram (ECG). Participant has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 50 to 90 mm Hg for diastolic, if out of range may be repeated once for eligibility determination at the Screening Visit or Check-in (Day -1 of Period 1).
18. Has a resting heart rate outside the range 50 to 90 beats per minute (bpm), if out of range may be repeated once for eligibility determination at the Screening Visit and/or Check-in (Day -1 of Period 1).
19. Has a QT interval with Fridericia correction method (QTcF) greater than (>) 430 milliseconds (ms) or PR outside the range 120 to 220 ms, if out of range may be repeated once for eligibility determination within a maximum of 5 minutes, at the Screening Visit and/or Check-in (Day -1 of Period 1).
20. Has abnormal Screening laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 upper limit of normal (ULN).
21. Has a history of Axis I/II mental disorders according to DSM-IV Axis I/II such as depression, anxiety disorders, bipolar disorder, attention deficit/hyperactivity disorder (ADHD), autism spectrum disorders, anorexia nervosa, bulimia nervosa, and schizophrenia.
22. Has a history of head injury or trauma.
23. Has any condition that would prevent an MRI from accurately or safely being performed (e.g., claustrophobia, cardiac pacemaker, metallic implants or clips), as verified per study site's standard MRI assessment questionnaire.
24. Has a risk of suicide according to the Investigator's clinical judgment (e.g., per Columbia-Suicide Severity Rating Scale [C-SSRS]) or has made a suicide attempt in the previous 6 months prior to Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Development Center Americas, Inc.
Locations (1):
- The Brain Institute, University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 27 June 2013 to 28 August 2014.
Pre-assignment Details: Healthy male participants were enrolled in this 3 period study and randomized in 1 of 9 administration sequences to receive TAK-063 3 mg, TAK-063 10 mg, TAK-063 30 mg and TAK-063 matching placebo. Due to predicted exposures being higher than likely clinically relevant, the dose of 300 mg was removed and replaced by 10 mg in protocol amendment 3.
Groups:
- Placebo + TAK-063 3 mg + TAK-063 30 mg: TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- TAK-063 3 mg + TAK-063 30 mg + Placebo: TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- TAK-063 30 mg + Placebo + TAK-063 3 mg: TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg: TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo: TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 placebo-matching tablets orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg: TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo: TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
- TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg: TAK-063 300 mg (participants enrolled before protocol amendment 3) or 10 mg (participants enrolled after protocol amendment 3), , tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of first intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 placebo-matching tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of second intervention period (1 day), followed by 7 days washout period, further followed by TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously once only on Day 1 of third intervention period (1 day).
Period: First Intervention Period (1 Day)
Arm/Group | Placebo + TAK-063 3 mg + TAK-063 30 mg | TAK-063 3 mg + TAK-063 30 mg + Placebo | TAK-063 30 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg | TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg | TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Placebo + TAK-063 3 mg + TAK-063 30 mg | TAK-063 3 mg + TAK-063 30 mg + Placebo | TAK-063 30 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg | TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg | TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Not Completed | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Noncompliance, Irritability | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Second Intervention Period (1 Day)
Arm/Group | Placebo + TAK-063 3 mg + TAK-063 30 mg | TAK-063 3 mg + TAK-063 30 mg + Placebo | TAK-063 30 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg | TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg | TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg
Started | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Completed | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Placebo + TAK-063 3 mg + TAK-063 30 mg | TAK-063 3 mg + TAK-063 30 mg + Placebo | TAK-063 30 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg | TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg | TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg
Started | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Completed | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period (1 Day)
Arm/Group | Placebo + TAK-063 3 mg + TAK-063 30 mg | TAK-063 3 mg + TAK-063 30 mg + Placebo | TAK-063 30 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg | TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg | TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg
Started | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Completed | 3 | 3 | 1 | 2 | 3 | 2 | 2 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set included all participants who were randomized to either 1 of the 9 treatment sequences.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + TAK-063 3 mg + TAK-063 30 mg | TAK-063 3 mg + TAK-063 30 mg + Placebo | TAK-063 30 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 3 mg + TAK-063 300 mg/10 mg | TAK-063 3 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 3 mg | Placebo + TAK-063 30 mg + TAK-063 300 mg/10 mg | TAK-063 30 mg + TAK-063 300 mg/10 mg + Placebo | TAK-063 300 mg/10 mg + Placebo + TAK-063 30 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (3.21) | 28.7 (7.64) | 23.7 (6.66) | 32.3 (5.13) | 23 (5.20) | 22.3 (3.51) | 27 (7.94) | 24.7 (2.08) | 23.7 (5.69) | 25.9 (5.60)
Sex/Gender, Customized [Number; unit: participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Non Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Pacific Islander-White | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 24
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 27
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 179 (2.65) | 182 (4.58) | 177 (8.19) | 187.7 (3.79) | 179.7 (10.79) | 182.3 (3.06) | 183.3 (8.14) | 183.3 (6.51) | 182.7 (4.51) | 181.9 (6.06)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 83.23 (11.981) | 93.80 (4.784) | 79.87 (16.910) | 82.3 (12.643) | 87.47 (13.955) | 77.33 (8.107) | 81.10 (5.821) | 86.40 (4.939) | 79.07 (11.716) | 83.40 (10.306)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.06 (4.430) | 28.38 (2.557) | 25.30 (3.190) | 23.39 (3.844) | 26.99 (2.108) | 23.28 (2.611) | 24.20 (2.417) | 25.71 (1.011) | 23.69 (3.269) | 25.22 (2.997)
Smoking Classification [Number; unit: participants]
  Never smoked | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 23
  Ex-smoker | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 4
Caffeine Consumption [Number; unit: participants]
  Consumes Caffiene | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 24
  Not consumes Caffiene | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Ketamine-Induced Brain Activity in Regions of Interest During Resting State
Description: Ketamine model was used to enhance the sensitivity to detect an effect of phosphodiesterase 10a (PDE10a) inhibition by TAK-063 by ketamine using neuroimaging battery tests. Ketamine induced robust blood oxygen level-dependent(BOLD) functional magnetic resonance imaging(fMRI) response while maintaining minimal accompanying psychotomimetic symptoms. The regions of interest include:left anterior cingulate cortex,right anterior cingulate cortex,left posterior cingulate cortex,right posterior cingulate cortex,left striatum,right striatum,left amygdala,right amygdala,left substantia nigra,right substantia nigra,left thalamus,right thalamus,left ventrolateral prefrontal cortex,right ventrolateral prefrontal cortex,left dorsolateral prefrontal cortex,right dorsolateral prefrontal cortex,left hippocampus,right hippocampus,left subgenual cingulate/Ba25,right subgenual cingulate/Ba25,left paracingulate gyrus/Ba32, and right paracingulate gyrus/Ba32.
Time Frame: Day 1: 4 hours post TAK-063 dose or placebo
Population: The pharmacodynamic (PD) analysis set included all participants in the safety set and with at least 1 valid PD assessment. PD analysis set did not include 2 participants treated with TAK-063 300 mg.
Measure: Mean (Standard Deviation); unit: percent signal change in brain activity
Groups:
- Placebo: TAK-063 placebo-matching tablets, orally and ketamine, infusion, intravenously on Day 1 in either intervention period 1, 2 or 3.
- TAK-063 3 mg: TAK-063 3 mg, tablets, orally along with ketamine, infusion, intravenously on Day 1 in either intervention period 1, 2 or 3.
- TAK-063 10 mg: TAK-063 10 mg, tablets, orally along with ketamine, infusion, intravenously on Day 1 in intervention period 1, 2 or 3.
- TAK-063 30 mg: TAK-063 30 mg, tablets, orally along with ketamine, infusion, intravenously on Day 1 in intervention period 1, 2 or 3.
Arm/Group | Placebo | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg
Number analyzed (Participants) | 22 | 14 | 14 | 15
percent signal change in brain activity
  Left Anterior Cingulate Cortex | 0.4954 (0.53382) | 0.2943 (0.67925) | 0.4439 (0.72261) | 0.3876 (0.47127)
  Right Anterior Cingulate Cortex | 0.4611 (0.44870) | 0.2542 (0.55542) | 0.4199 (0.70069) | 0.3251 (0.47592)
  Left Posterior Cingulate Cortex | 0.4922 (0.52563) | 0.4647 (0.52746) | 0.5316 (0.77685) | 0.3987 (0.49018)
  Right Posterior Cingulate Cortex | 0.5412 (0.52336) | 0.4515 (0.57054) | 0.6132 (0.79296) | 0.3783 (0.55473)
  Left Striatum | 0.2914 (0.40513) | 0.0644 (0.47601) | 0.3045 (0.51442) | 0.2453 (0.40828)
  Right Striatum | 0.3605 (0.37202) | 0.1154 (0.52174) | 0.3124 (0.46817) | 0.2617 (0.36033)
  Left Amygdala | 0.3413 (0.66866) | 0.4776 (0.72631) | 0.4888 (0.60449) | 0.3435 (0.57560)
  Right Amygdala | 0.2102 (0.72431) | 0.1180 (0.85125) | 0.0106 (0.76838) | 0.2686 (0.53395)
  Left Substantia Nigra | 0.3989 (0.49787) | 0.2857 (0.61851) | 0.5560 (0.67716) | 0.2214 (0.36486)
  Right Substantia Nigra | 0.2925 (0.45514) | 0.2209 (0.69383) | 0.3398 (0.45331) | 0.1148 (0.40258)
  Left Thalamus | 0.5166 (0.40051) | 0.3406 (0.58293) | 0.5564 (0.52695) | 0.3589 (0.43768)
  Right Thalamus | 0.4807 (0.35272) | 0.3392 (0.59598) | 0.5159 (0.44482) | 0.3734 (0.44173)
  Left Ventrolateral Prefrontal Cortex | 0.6355 (0.79768) | 0.5183 (0.66695) | 0.6081 (0.73306) | 0.5900 (0.47920)
  Right Ventrolateral Prefrontal Cortex | 0.7932 (0.59179) | 0.5134 (0.69396) | 0.6661 (0.75274) | 0.6119 (0.44821)
  Left Dorsolateral Prefrontal Cortex | 0.3918 (0.41983) | 0.2576 (0.56173) | 0.4451 (0.62506) | 0.3720 (0.30576)
  Right Dorsolateral Prefrontal Cortex | 0.4715 (0.40803) | 0.2799 (0.53268) | 0.5403 (0.78105) | 0.4331 (0.39160)
  Left Hippocampus | 0.3150 (0.37531) | 0.1790 (0.47311) | 0.3073 (0.41116) | 0.2123 (0.35146)
  Right Hippocampus | 0.2540 (0.27489) | 0.1814 (0.51038) | 0.2141 (0.34537) | 0.0989 (0.35725)
  Left Subgenual Cingulate/BA25 | -0.3974 (1.60367) | 0.2236 (1.22450) | -0.2448 (1.46965) | -0.0002 (2.18015)
  Right Subgenual Cingulate/BA25 | -0.1463 (1.55680) | -0.3430 (1.15319) | -0.6379 (2.30349) | 0.0424 (1.71727)
  Left Paracingulate Gyrus/BA32 | 0.4776 (0.43067) | 0.2799 (0.59577) | 0.4069 (0.65537) | 0.3281 (0.38990)
  Right Paracingulate Gyrus/BA32 | 0.5849 (0.51897) | 0.3583 (0.58987) | 0.4972 (0.82842) | 0.3969 (0.52267)
Statistical Analysis 1: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Anterior Cingulate Cortex: Values were obtained using analysis of variance (ANOVA) model with sequence, period, regimen and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.259, ANOVA; Least Squares (LS) Mean Difference = -0.2348, 95% CI 2-sided [-0.6506 to 0.1809], Standard Error of Mean 0.20458 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 2: Comparison: Placebo vs TAK-063 10 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Anterior Cingulate Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.869, ANOVA; LS Mean Difference = -0.0367, 95% CI 2-sided [-0.4853 to 0.4119], Standard Error of Mean 0.22075 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 3: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.306, ANOVA; LS Mean Difference = -0.2180, 95% CI 2-sided [-0.6441 to 0.2081], Standard Error of Mean 0.20968 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 4: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Anterior Cingulate Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.169, ANOVA; LS Mean Difference = -0.2525, 95% CI 2-sided [-0.6174 to 0.1124], Standard Error of Mean 0.17956 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 5: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.831, ANOVA; LS Mean Difference = -0.0417, 95% CI 2-sided [-0.4354 to 0.3521], Standard Error of Mean 0.19375 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 6: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.197, ANOVA; LS Mean Difference = -0.2421, 95% CI 2-sided [-0.6161 to 0.1319], Standard Error of Mean 0.18403 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 7: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Posterior Cingulate Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.480, ANOVA; LS Mean Difference = -0.1155, 95% CI 2-sided [-0.4443 to 0.2133], Standard Error of Mean 0.16180 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 8: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p = 0.345, ANOVA; LS Mean Difference = 0.1673, 95% CI 2-sided [-0.1875 to 0.5221], Standard Error of Mean 0.17458 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 9: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p = 0.371, ANOVA; LS Mean Difference = -0.1504, 95% CI 2-sided [-0.4874 to 0.1866], Standard Error of Mean 0.16583 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 10: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Posterior Cingulate Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.364, ANOVA; LS Mean Difference = -0.1731, 95% CI 2-sided [-0.5553 to 0.2092], Standard Error of Mean 0.18808 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 11: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; p = 0.507, ANOVA; LS Mean Difference = 0.1362, 95% CI 2-sided [-0.2762 to 0.5486], Standard Error of Mean 0.20294 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 12: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; p = 0.210, ANOVA; LS Mean Difference = -0.2464, 95% CI 2-sided [-0.6381 to 0.1453], Standard Error of Mean 0.19276 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 13: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Striatum: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.039, ANOVA; LS Mean Difference = -0.3059, 95% CI 2-sided [-0.5955 to -0.0162], Standard Error of Mean 0.14253 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 14: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.931, ANOVA; LS Mean Difference = 0.0134, 95% CI 2-sided [-0.2991 to 0.3260], Standard Error of Mean 0.15380 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 15: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.431, ANOVA; LS Mean Difference = -0.1164, 95% CI 2-sided [-0.4133 to 0.1804], Standard Error of Mean 0.14608 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 16: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Striatum: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.020, ANOVA; LS Mean Difference = -0.3269, 95% CI 2-sided [-0.5985 to -0.0554], Standard Error of Mean 0.13362 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 17: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; p = 0.562, ANOVA; LS Mean Difference = -0.0845, 95% CI 2-sided [-0.3775 to 0.2085], Standard Error of Mean 0.14418 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 18: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; p = 0.216, ANOVA; LS Mean Difference = -0.1727, 95% CI 2-sided [-0.4510 to 0.1056], Standard Error of Mean 0.13695 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 19: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Amygdala: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.962, ANOVA; LS Mean Difference = -0.0084, 95% CI 2-sided [-0.3663 to 0.3495], Standard Error of Mean 0.17609 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 20: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 19]; Test type: Superiority or Other; p = 0.852, ANOVA; LS Mean Difference = -0.0357, 95% CI 2-sided [-0.4218 to 0.3505], Standard Error of Mean 0.19001 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 21: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 19]; Test type: Superiority or Other; p = 0.241, ANOVA; LS Mean Difference = -0.2154, 95% CI 2-sided [-0.5822 to 0.1514], Standard Error of Mean 0.18048 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 22: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Amygdala: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.443, ANOVA; LS Mean Difference = -0.1380, 95% CI 2-sided [-0.4991 to 0.2230], Standard Error of Mean 0.17766 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 23: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 22]; Test type: Superiority or Other; p = 0.295, ANOVA; LS Mean Difference = -0.2037, 95% CI 2-sided [-0.5933 to 0.1859], Standard Error of Mean 0.19170 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 24: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 22]; Test type: Superiority or Other; p = 0.743, ANOVA; LS Mean Difference = -0.0602, 95% CI 2-sided [-0.4303 to 0.3098], Standard Error of Mean 0.18209 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 25: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Substantia Nigra: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.277, ANOVA; LS Mean Difference = -0.1774, 95% CI [-0.5040 to 0.1491], Standard Error of Mean 0.16068 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 26: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.758, ANOVA; LS Mean Difference = -0.0539, 95% CI 2-sided [-0.4062 to 0.2985], Standard Error of Mean 0.17338 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 27: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.012, ANOVA; LS Mean Difference = -0.4377, 95% CI 2-sided [-0.7724 to -0.1031], Standard Error of Mean 0.16468 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 28: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Substantia Nigra: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.490, ANOVA; LS Mean Difference = -0.1037, 95% CI 2-sided [-0.4055 to 0.1981], Standard Error of Mean 0.14849 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 29: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.534, ANOVA; LS Mean Difference = -0.1007, 95% CI 2-sided [-0.4263 to 0.2249], Standard Error of Mean 0.16023 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 30: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.169, ANOVA; LS Mean Difference = -0.2140, 95% CI 2-sided [-0.5233 to 0.0953], Standard Error of Mean 0.15219 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 31: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Thalamus: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.070, ANOVA; LS Mean Difference = -0.2641, 95% CI 2-sided [-0.5510 to 0.0228], Standard Error of Mean 0.14118 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 32: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.579, ANOVA; LS Mean Difference = -0.0854, 95% CI 2-sided [-0.3950 to 0.2242], Standard Error of Mean 0.15234 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 33: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.100, ANOVA; LS Mean Difference = -0.2446, 95% CI 2-sided [-0.5387 to 0.0494], Standard Error of Mean 0.14470 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 34: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Thalamus: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.113, ANOVA; LS Mean Difference = -0.2200, 95% CI 2-sided [-0.4950 to 0.0550], Standard Error of Mean 0.13533 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 35: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.720, ANOVA; LS Mean Difference = -0.0527, 95% CI 2-sided [-0.3495 to 0.2440], Standard Error of Mean 0.14603 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 36: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.196, ANOVA; LS Mean Difference = -0.1830, 95% CI 2-sided [-0.4649 to 0.0989], Standard Error of Mean 0.13870 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 37: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Ventrolateral Prefrontal Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.313, ANOVA; LS Mean Difference = -0.2051, 95% CI 2-sided [-0.6122 to 0.2020], Standard Error of Mean 0.20032 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 38: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.908, ANOVA; LS Mean Difference = 0.0253, 95% CI 2-sided [-0.4140 to 0.4646], Standard Error of Mean 0.21616 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 39: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.148, ANOVA; LS Mean Difference = -0.3042, 95% CI 2-sided [-0.7214 to 0.1131], Standard Error of Mean 0.20531 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 40: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Ventrolateral Prefrontal Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.067, ANOVA; LS Mean Difference = -0.3409, 95% CI 2-sided [-0.7066 to 0.0249], Standard Error of Mean 0.17997 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 41: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.739, ANOVA; LS Mean Difference = -0.0652, 95% CI 2-sided [-0.4599 to 0.3294], Standard Error of Mean 0.19419 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 42: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean Difference = -0.4163, 95% CI 2-sided [-0.7912 to -0.0415], Standard Error of Mean 0.18445 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 43: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Dorsolateral Prefrontal Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.166, ANOVA; LS Mean Difference = -0.2032, 95% CI 2-sided [-0.4952 to 0.0888], Standard Error of Mean 0.14369 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 44: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.552, ANOVA; LS Mean Difference = 0.0932, 95% CI 2-sided [-0.2219 to 0.4083], Standard Error of Mean 0.15504 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 45: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.271, ANOVA; LS Mean Difference = -0.1648, 95% CI 2-sided [-0.4641 to 0.1345], Standard Error of Mean 0.14727 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 46: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Dorsolateral Prefrontal Cortex: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.129, ANOVA; LS Mean Difference = -0.2516, 95% CI 2-sided [-0.5802 to 0.0770], Standard Error of Mean 0.16169 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 47: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 46]; Test type: Superiority or Other; p = 0.468, ANOVA; LS Mean Difference = 0.1279, 95% CI 2-sided [-0.2266 to 0.4825], Standard Error of Mean 0.17447 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 48: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 46]; Test type: Superiority or Other; p = 0.228, ANOVA; LS Mean Difference = -0.2033, 95% CI 2-sided [-0.5401 to 0.1334], Standard Error of Mean 0.16572 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 49: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Hippocampus: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.141, ANOVA; LS Mean Difference = -0.2000, 95% CI 2-sided [-0.4696 to 0.0696], Standard Error of Mean 0.13268 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 50: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 49]; Test type: Superiority or Other; p = 0.964, ANOVA; LS Mean Difference = -0.0065, 95% CI 2-sided [-0.2975 to 0.2844], Standard Error of Mean 0.14317 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 51: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 49]; Test type: Superiority or Other; p = 0.164, ANOVA; LS Mean Difference = -0.1935, 95% CI 2-sided [-0.4699 to 0.0828], Standard Error of Mean 0.13599 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 52: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Hippocampus: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.285, ANOVA; LS Mean Difference = -0.1446, 95% CI 2-sided [-0.4152 to 0.1260], Standard Error of Mean 0.13315 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 53: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 52]; Test type: Superiority or Other; p = 0.903, ANOVA; LS Mean Difference = -0.0176, 95% CI 2-sided [-0.3096 to 0.2744], Standard Error of Mean 0.14368 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 54: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 52]; Test type: Superiority or Other; p = 0.245, ANOVA; LS Mean Difference = -0.1615, 95% CI 2-sided [-0.4388 to 0.1159], Standard Error of Mean 0.13647 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 55: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Subgenual Cingulate/BA25: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.429, ANOVA; LS Mean Difference = 0.3659, 95% CI 2-sided [-0.5630 to 1.2948], Standard Error of Mean 0.45708 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 56: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 55]; Test type: Superiority or Other; p = 0.937, ANOVA; LS Mean Difference = 0.0395, 95% CI 2-sided [-0.9628 to 1.0419], Standard Error of Mean 0.49321 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 57: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 55]; Test type: Superiority or Other; p = 0.101, ANOVA; LS Mean Difference = 0.7902, 95% CI 2-sided [-0.1618 to 1.7423], Standard Error of Mean 0.46847 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 58: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Subgenual Cingulate/BA25: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.321, ANOVA; LS Mean Difference = -0.4404, 95% CI 2-sided [-1.3296 to 0.4488], Standard Error of Mean 0.43756 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 59: Comparison: Placebo vs TAK-063 10 mg; [analysis description as in outcome 1, analysis 58]; Test type: Superiority or Other; p = 0.328, ANOVA; LS Mean Difference = -0.4685, 95% CI 2-sided [-1.4280 to 0.4910], Standard Error of Mean 0.47214 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 60: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 58]; Test type: Superiority or Other; p = 0.356, ANOVA; LS Mean Difference = 0.4200, 95% CI 2-sided [-0.4914 to 1.3314], Standard Error of Mean 0.44846 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 61: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Paracingulte gyrus/BA32. Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.188, ANOVA; LS Mean Difference = -0.2254, 95% CI 2-sided [-0.5666 to 0.1158], Standard Error of Mean 0.16790 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 62: Comparison: Placebo vs TAK-063 10 mg; Test the equality on the means between TAK-063 and Placebo for the region Left Paracingulte gyrus/BA32: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.899, ANOVA; LS Mean Difference = -0.0232, 95% CI 2-sided [-0.3914 to 0.3449], Standard Error of Mean 0.18117 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 63: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 62]; Test type: Superiority or Other; p = 0.150, ANOVA; LS Mean Difference = -0.2534, 95% CI 2-sided [-0.6032 to 0.0963], Standard Error of Mean 0.17208 — Difference between least square means of TAK-063 30 mg and Placebo
Statistical Analysis 64: Comparison: Placebo vs TAK-063 3 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Paracingulte gyrus/BA3: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.148, ANOVA; LS Mean Difference = -0.2821, 95% CI 2-sided [-0.6690 to 0.1048], Standard Error of Mean 0.19038 — Difference between least square means of TAK-063 3 mg and Placebo
Statistical Analysis 65: Comparison: Placebo vs TAK-063 10 mg; Test the equality on the means between TAK-063 and Placebo for the region Right Paracingulte gyrus/BA32: Values were obtained using an ANOVA model with sequence, period, regimen, and participant nested within sequence as factors by regions of interest; Test type: Superiority or Other; p = 0.817, ANOVA; LS Mean Difference = -0.0480, 95% CI 2-sided [-0.4655 to 0.3695], Standard Error of Mean 0.20543 — Difference between least square means of TAK-063 10 mg and Placebo
Statistical Analysis 66: Comparison: Placebo vs TAK-063 30 mg; [analysis description as in outcome 1, analysis 65]; Test type: Superiority or Other; p = 0.091, ANOVA; LS Mean Difference = -0.3395, 95% CI 2-sided [-0.7361 to 0.0570], Standard Error of Mean 0.19513 — Difference between least square means of TAK-063 30 mg and Placebo

2. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-063 and TAK-063 Metabolite (M-I)
Time Frame: Day 1: pre-dose and at multiple time points (up to 24 hours) postdose
Population: The pharmacokinetic (PK) analysis set included all participants in the safety set and with at least 1 measurable plasma concentration. PK analysis set did not include 2 participants treated with 300 mg.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg
Number analyzed (Participants) | 14 | 14 | 15
nanogram per milliliter (ng/mL)
  TAK-063 | 10.35 (2.860) [0.5 to 6.0] | 48.16 (8.769) | 109.9 (27.053)
  M-I | 12.07 (3.235) | 48.94 (11.500) | 103.72 (32.635)

3. Secondary Outcome: Tmax: Time to Reach Cmax for TAK-063 and TAK-063 M-I
Time Frame: Day 1: pre-dose and at multiple time points (up to 24 hours) postdose
Population: The PK analysis set included all participants in the safety set and with at least 1 measurable plasma concentration. PK analysis set did not include 2 participants treated with 300 mg.
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg
Number analyzed (Participants) | 14 | 14 | 15
hours
  TAK-063 | 3.02 (2.860) [0.5 to 6.0] | 3.03 [2.0 to 5.8] | 3.02 [2.0 to 5.8]
  M-I | 2.96 [1.9 to 4.3] | 3.03 [2.0 to 5.7] | 4.23 [2.0 to 6.0]

4. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-063 and TAK-063 M-I
Time Frame: Day 1: Pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg
Number analyzed (Participants) | 14 | 14 | 15
nanogram hours per milliliter (ng*hr/mL)
  TAK-063 | 111.36 (38.460) | 548.58 (122.686) | 1298.89 (331.095)
  M-I | 114.81 (48.453) | 582.91 (201.503) | 1285.18 (499.431)

5. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to 14 days after last dose of study drug (Day 32)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- TAK-063 300 mg: TAK-063 300 mg, tablets, orally along with ketamine, infusion, intravenously on Day 1 in intervention period 1, 2 and 3.
Arm/Group | Placebo | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg | TAK-063 300 mg
Number analyzed (Participants) | 22 | 14 | 14 | 15 | 2
percentage of participants | 68.2 | 50 | 57.1 | 86.7 | 100

6. Secondary Outcome: Percentage of Participants Who Meet the Takeda Global Research and Development Center, Inc. (TGRD) Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Description: The percentage of participants with any markedly abnormal standard safety laboratory values collected throughout study.
Time Frame: Baseline up to 14 days after last dose of study drug (Day 32)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg | TAK-063 300 mg
Number analyzed (Participants) | 22 | 14 | 14 | 15 | 2
percentage of participants | 9.1 | 0 | 14.3 | 6.7 | 0

7. Secondary Outcome: Percentage of Participants Who Meet the TGRD Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Description: The percentage of participants who meet markedly abnormal criteria designated by TGRD. Vital signs included oral temperature, respiration, blood pressure and pulse (beats per minute).
Time Frame: Baseline up to 14 days after last dose of study drug (Day 32)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg | TAK-063 300 mg
Number analyzed (Participants) | 22 | 14 | 14 | 15 | 2
percentage of participants | 50.0 | 64.3 | 57.1 | 53.3 | 100

8. Secondary Outcome: Percentage of Participants Who Meet the TGRD Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post Dose
Description: The percentage of participants who meet markedly abnormal criteria designated by TGRD measured throughout study.
Time Frame: Baseline up to 14 days after last dose of study drug (Day 32)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg | TAK-063 300 mg
Number analyzed (Participants) | 22 | 14 | 14 | 15 | 2
percentage of participants | 27.3 | 14.3 | 35.7 | 53.3 | 100

ADVERSE EVENTS:
Time Frame: Baseline up to 14 days after last dose of study drug (Day 32)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-063 3 mg | TAK-063 10 mg | TAK-063 30 mg | TAK-063 300 mg
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/14 | 0/14 | 0/15 | 0/2
Other Adverse Events (participants affected / at risk) | 15/22 | 7/14 | 8/14 | 13/15 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | TAK-063 3 mg (N=14) | TAK-063 10 mg (N=14) | TAK-063 30 mg (N=15) | TAK-063 300 mg (N=2)
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 3 | 6 | 8 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 3 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 4 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 4 | 7 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Coordination Abnormal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 2 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Communication Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 3 | 2 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property